CLINICAL TRIAL: NCT02558660
Title: Evaluating Use of a Farmers Market Incentive Program Among Low-Income Health Center Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Alicia Cohen, Clinical Lecturer, Robert Wood Johnson Foundation Clinical Scholar, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HUM00076630
Record Dates: First submitted 2015-09-04; First posted 2015-09-24 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Food Insecurity; Non-use of Existing State-wide SNAP Incentive Program
Keywords: Supplemental Nutrition Incentive Program (SNAP); economic incentive
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Double Up Food Bucks (Experimental): Clinic-based educational intervention about an existing SNAP healthy food incentive program, as well as a $10 voucher to spend on produce at farmers markets
  Interventions: Behavioral: Education; Behavioral: voucher

INTERVENTIONS:
Behavioral: Education — Educational intervention about an existing SNAP healthy food incentive program
Behavioral: voucher — $10 voucher to spend on produce at farmers markets

SUMMARY:
The purpose of this study is to evaluate the impact of a brief clinic-based educational intervention on utilization of Double Up Food Bucks (DUFB)-a Michigan-wide Supplemental Nutrition Assistance Program (SNAP) healthy food incentive--among low income health center patients at a community health center in Southeast Michigan.

DETAILED DESCRIPTION:
Study participants were provided a 3-5 minute explanation of DUFB, written program materials, and initial $10 market voucher. Participants were surveyed four times over five months, and a subset are also participating in post-intervention focus groups.

ELIGIBILITY:
Inclusion Criteria:

* patient or family member of patient
* at least 18 years of age
* currently SNAP-enrolled
* identifies as one of primary food shoppers for household
* English or Spanish-speaking

Exclusion Criteria:

* under 18
* not currently SNAP-enrolled
* not one of primary food shoppers for household
* unable to complete a telephone survey in English or Spanish
* unable to provide a working telephone number where they could be contacted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of participant DUFB use over time, as assessed by an interviewer-administered survey using structured open-ended questions | 5 months
  Use of DUFB at baseline assessed with yes/no response. At each of the the 3 follow-up surveys waves (1.5 months, 3 months, and 5 months), participants will be asked if they have used DUFB in the past month (yes/no), and if yes, how many times.
Participant-perceived barriers and facilitators to DUFB use following educational intervention, as assessed by an interviewer-administered survey using structured open-ended questions and semi-structured focus group questions | 12 months
  Through an iterative process, three team members will independently conduct thematic analyses, compared codes, resolve discrepancies, and summarize key thematic findings.

SECONDARY OUTCOMES:
Change from baseline fruit and vegetable consumption at 1.5 months, 3 months, and 5 months, as assessed by a validated 2 question fruit and vegetable screener | baseline, 1.5 months, 3 months, 5 months
  Servings/day range from 0 to >=4 (scale applied separately to fruit consumption and vegetable consumption. Change will be calculated from two time points at each of three follow-up periods (1.5 months, 3 months, and 5 months) minus the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Cohen, MD, Principal Investigator — University of Michigan
Locations (1):
- Ypsilanti Health Center, University of Michigan, Ypsilanti, Michigan, United States